CLINICAL TRIAL: NCT05215860
Title: Visual Communication Through Personal Intraoral Photographs of Oral Potentially Malignant Disorders in Current Tobacco and Areca Nut Users Improves Habit Abstinence: a Pilot Interventional Study
Brief Title: Photographic Evidence of Oral Precancerous Lesions in Current Tobacco and Areca Nut Users Improves Their Quit Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Shalini Gupta, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IEC-616
Record Dates: First submitted 2021-12-25; First posted 2022-01-31 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Precancerous Conditions
Keywords: cessation; tobacco use; smokeless tobacco; areca; intraoral photography; abstinence
MeSH Terms: conditions — Precancerous Conditions; Tobacco Use | interventions — Tobacco Products

STUDY DESIGN:
Intervention Model Description: A prospective pilot interventional longitudinal study
Who Masked: Investigator
Masking Description: The investigator who provided behavioural counselling to the participants was blinded to their clinical diagnosis of oral lesions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habit cessation counselling with management for OPMD (Active Comparator): n=100; Habit cessation counselling with general and medical management for OPMD
  Interventions: Behavioral: Tobacco and areca nut cessation counselling with standard management for Oral Potentially Malignant Disorders
- Habit cessation counselling, management for OPMD and intraoral photographs (Experimental): n=100; Habit cessation counselling with standard management for OPMD and visual exposure to personal intraoral photographs of oral lesions at baseline and review
  Interventions: Behavioral: Tobacco and areca nut cessation counselling with standard management for Oral Potentially Malignant Disorders; Other: visual exposure to personal intraoral photographs of oral lesions at baseline and review

INTERVENTIONS:
Behavioral: Tobacco and areca nut cessation counselling with standard management for Oral Potentially Malignant Disorders — WHO toolkit for Tobacco cessation (5A's and 5R's model)
Other: visual exposure to personal intraoral photographs of oral lesions at baseline and review — Chairside digital intraoral photographs of oral potentially malignant disorder with smart phone and showing the photograph to the participant explaining the abnormal areas of concern
  Arms: Habit cessation counselling, management for OPMD and intraoral photographs

SUMMARY:
The success of tobacco and areca nut cessation programs in individuals with Oral Potentially Malignant Disorders (OPMDs) is imperative for risk reduction and prevention of oral cancer. A prospective pilot interventional study where 200 participants with current tobacco and areca nut habits and OPMD were randomly divided in two groups. Group A ( n=100; Habit cessation counselling with general and medical management for OPMD). Group B ( n=100; Habit cessation counselling with general and medical management for OPMD and visual exposure to personal intraoral photographs of oral lesions at baseline and review).

DETAILED DESCRIPTION:
A prospective pilot interventional study was carried out in a Oral Medicine unit at a tertiary referral center where OPMD and Oral cancer screening is carried out routinely in all patients examined in the Out Patient Department (OPD). Ethical clearance for conducting the study and taking serial intraoral photographs of OPMD in consenting participants was obtained from the Institute Ethics Committee.All patients in OPD were initially screened for current habits of any form of tobacco and areca nut products through history and referred to the Tobacco Cessation Clinic (TCC) for individual counselling session.This counselling was based on the toolkit issued by the World Health Organization (WHO) for delivering brief tobacco intervention under WHO capacity building training package.The patients then underwent detailed intraoral examination for any oral mucosal changes. Those patients that were diagnosed as having any OPMD as per clinical diagnostic criteria were then recruited as participants in the study. A total of 200 participants with current tobacco and areca nut habits and OPMDs were recruited after informed written consent and randomly assigned to the two groups. The Control Group A had 100 participants who received standard management protocol for OPMD. The experimental Group B received all the management as in Control Group A but were also shown their intraoral photographs of oral lesions and explained about the areas of abnormalities that were of concern. All the participants were reviewed at 1, 3 and 6 months for surveillance of OPMD lesions and habit status.The data was analysed for statistically significant differences between the two groups p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Current tobacco and areca nut users.
* Presence of oral potentially malignant disorders

Exclusion Criteria:

• Any oral lesion suspicious of malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Habit quit rates | 6 months
  Discontinuation of habit more than 1 month.

SECONDARY OUTCOMES:
Size of oral lesions | 6 months
  Change in size of lesions from baseline in millimeters
Oral burning sensation | 6 months
  Change in oral burning sensation from baseline Visual Analogue Scale (VAS) scale 0-10; 0: No oral burning sensation; 10: Worst oral burning sensation
Colour of oral lesions | 6 months
  Change in colour of oral lesions from red to white
Inter incisal mouth opening | 6 months
  Change in interincisal mouth opening from baseline in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Gupta, MDS,FDSRCS, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Oral Medicine and Radiology, CDER, AIIMS, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
The study data can be made available on request via email to principal investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after publication in journal for a period of 12 months
Access Criteria: email of principal investigator shalinigupta@hotmail.com